CLINICAL TRIAL: NCT07242339
Title: Comparison of the Analgesic Efficacy of Adductor Canal Block Versus Adductor Canal Plus Biceps Femoris Short Head Block in Patients Undergoing Knee Arthroscopy: A Prospective Randomized Controlled Trial
Brief Title: Comparison of the Analgesic Efficacy of Adductor Canal Block Versus Adductor Canal Plus Biceps Femoris Short Head Block in Patients Undergoing Knee Arthroscopy
Acronym: bifes knee
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kanuni Sultan Suleyman Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Engin Ihsan Turan, principal investigator, Kanuni Sultan Suleyman Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: Bifes knee
Record Dates: First submitted 2025-11-17; First posted 2025-11-21 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2025-11

CONDITIONS: Postoperative Pain Management
Keywords: regional anesthesia
MeSH Terms: interventions — Single Person

STUDY DESIGN:
Intervention Model Description: Participants will be randomized in a 1:1 ratio to receive either an adductor canal block (ACB) or a combined adductor canal plus biceps femoris short head (ACB+BiFeS) block. Both interventions will be performed under ultrasound guidance at the end of surgery.
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants will be blinded to group allocation. Outcome assessors recording pain scores, opioid consumption, and side effects will be blinded to the intervention. The anesthesiologists performing the blocks cannot be blinded due to the nature of the procedures.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Adductor Canal Block (ACB) (Active Comparator): Participants will undergo ultrasound-guided adductor canal block at the end of surgery under spinal anesthesia.
  Interventions: Procedure: Adductor Canal Block (ACB) Only
- Adductor Canal Block + Biceps Femoris Short Head Block (ACB+BiFeS) (Active Comparator): Participants will undergo both adductor canal block and biceps femoris short head block at the end of surgery under spinal anesthesia.
  Interventions: Procedure: biceps femoris short head block + Adductor Canal Block (ACB)

INTERVENTIONS:
Procedure: Adductor Canal Block (ACB) Only — Ultrasound-guided injection of 10 mL 0.25% bupivacaine into the adductor canal targeting the femoral artery region, providing motor-sparing analgesia to the medial/anterior knee.
  Arms: Adductor Canal Block (ACB)
Procedure: biceps femoris short head block + Adductor Canal Block (ACB) — Combination of adductor canal block (10 mL 0.25% bupivacaine) and biceps femoris short head block with 25 mL 0.25% bupivacaine, deposited at the interfascial plane between BiFeS muscle and lateral femoral cortex to extend analgesia to the posterolateral knee.
  Arms: Adductor Canal Block + Biceps Femoris Short Head Block (ACB+BiFeS)

SUMMARY:
This prospective, randomized, controlled, and multicenter clinical study aims to compare the postoperative analgesic efficacy of two regional anesthesia techniques commonly used in knee arthroscopy: adductor canal block (ACB) and combined adductor canal block plus biceps femoris short head (ACB+BiFeS) block. The study will evaluate postoperative pain control, opioid consumption, adverse effects, hospital stay, and patient satisfaction. Findings will help determine the most effective and safe method for postoperative analgesia in knee arthroscopy patients.

DETAILED DESCRIPTION:
Knee arthroscopy is one of the most common orthopedic procedures and is frequently associated with significant postoperative pain. Effective multimodal analgesia is therefore essential to reduce opioid consumption, improve early mobilization, and enhance overall patient recovery. Among the regional anesthesia techniques, the adductor canal block (ACB) is well established as an effective motor-sparing block that provides analgesia to the medial and anterior aspects of the knee. However, patients often continue to experience posterolateral knee pain, which is not consistently relieved by ACB alone.

Recent anatomical and cadaveric studies have described the biceps femoris short head (BiFeS) block as a promising technique for targeting the posterolateral knee compartment. The BiFeS block involves deposition of local anesthetic between the short head of the biceps femoris muscle and the lateral femoral cortex at the supracondylar level. Preliminary findings suggest that this block may provide effective analgesia for the posterolateral knee without causing significant motor impairment.

This prospective, randomized, controlled, multicenter clinical trial is designed to evaluate whether the addition of the BiFeS block to standard ACB improves postoperative analgesia compared with ACB alone in patients undergoing knee arthroscopy under spinal anesthesia. The study will investigate pain scores at rest and during movement, total opioid consumption, side effects, rescue analgesic requirements, and quality of recovery. The dermatomal distribution of the blocks will be optionally assessed using cold testing.

By directly comparing ACB and combined ACB+BiFeS block under standardized perioperative conditions, this study seeks to generate high-quality evidence on the clinical utility of BiFeS as an adjunct technique. The results are expected to guide anesthesiologists in selecting optimal regional analgesia strategies for knee arthroscopy, with the potential to improve patient satisfaction, reduce opioid-related complications, and shorten hospitalization.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* ASA physical status I-III
* Scheduled for elective knee arthroscopy under spinal anesthesia
* Ability to provide written informed consent

Exclusion Criteria:

* Coagulopathy or bleeding diathesis
* Current use of anticoagulant therapy
* Known allergy or contraindication to local anesthetics used in the study
* History of diabetes mellitus with neuropathy or other neuropathic disorders
* Contraindications to regional anesthesia techniques
* Refusal to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-11-20 (Actual); Primary Completion 2026-03-10 (Estimated); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
Total Opioid Consumption (Tramadol, mg) | 24 hours
  The total dose of tramadol administered via intravenous patient-controlled analgesia (PCA) device within the first 24 hours postoperatively will be recorded in milligrams.

SECONDARY OUTCOMES:
Postoperative Pain with Movement and at rest (NRS) | At 0, 6, 12, and 24 hours after surgery
  Pain intensity during knee movement will be assessed using the Numerical Rating Scale (0-10).
Rescue Analgesia Requirement | Within the first 24 hours postoperatively
  The number of patients requiring rescue analgesia (IV dexketoprofen 50 mg) will be recorded.
Incidence of Nausea and Vomiting | Within the first 24 hours postoperatively
  Presence of nausea/vomiting and the requirement for antiemetic medications will be documented.
Quality of Recovery (QOR-15 score) | At 24 hours after surgery
  Patient recovery quality will be assessed using the validated Quality of Recovery 15-item questionnaire (QOR-15). The scale includes 15 items, each scored from 0 to 10, producing a total score ranging from 0 to 150.
  Minimum score: 0 (poor recovery)
  Maximum score: 150 (excellent recovery)
  Interpretation: Higher scores indicate better postoperative recovery.
Dermatomal Spread of Block | 2nd hour postoperatively
  Sensory block distribution will be assessed using a cold test to map dermatomal coverage.
Motor Blockade Incidence | Within the first 24 hours postoperatively
  Patients will be evaluated for presence or absence of motor weakness attributable to the block.

CONTACTS AND LOCATIONS:
Overall Officials: Engin ihsan Turan, Specialist, Principal Investigator — Health Science University İstanbul Kanuni Sultan Süleyman Education and Training Hospital
Locations (1):
- Health Science University İstanbul Kanuni Sultan Süleyman Education and Training Hospital, Istanbul, küçükçekmece, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No